CLINICAL TRIAL: NCT03982836
Title: Impact of Different Dietary Fibers in Gastric Emptying Time and Intestinal Transit of Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, Principal Investigator, Federal University of Minas Gerais
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CAAE: 85797918.1.0000.5149
Record Dates: First submitted 2019-05-21; First posted 2019-06-12 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Gastric Emptying; Intestinal Transit Time
Keywords: Gastric Emptying; Scintigraphy; Intestinal Transit Time; Prebiotic; Soluble Dietary Fiber; Technetium-99m
MeSH Terms: interventions — Prebiotics

STUDY DESIGN:
Intervention Model Description: It is a cross-sectional study, where the volunteer should attend the study area on three different days with a minimum washout of 7 days, each day receiving a sandwich containing one of the modules studied in a randomized manner (Partially Hydrolyzed Guar Gum, Fructooligosaccharide or Maltodextrin) and will be instructed to ingest this sandwich in the maximum time of 10 minutes. The volunteers should on an 8-hour fast. Samples of blood will be collected in the fasting, 60 and 180 minutes after the injection of the sandwich for intestinal hormone dosage.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All subjects involved with this study will be masked. The masking was revealed only after the analysis of the results obtained.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fructooligosaccharide (Experimental): All the 25 volunteers received the sandwich containing 20 grams of fructooligosaccharide
  Interventions: Dietary Supplement: Soluble Dietary Fibers
- Partially hydrolyzed guar gum (Experimental): All the 25 volunteers received the sandwich containing 20 grams of partially hydrolyzed guar gum
  Interventions: Dietary Supplement: Soluble Dietary Fibers
- Maltodextrin (Placebo Comparator): All the 25 volunteers received the sandwich containing 20 grams of Maltodextrin
  Interventions: Dietary Supplement: Soluble Dietary Fibers

INTERVENTIONS:
Dietary Supplement: Soluble Dietary Fibers — All 25 volunteers received, were separated for 7 days of washout, one containing maltodextrin (control), Frutooligossacharide or guar gum partially hydrolyzed in a randomized manner. As the partially hydrolyzed guar gum and fructooligosaccharide, soluble dietary fibers that present different behaviors in the body.
  Other Names: Prebiotic; Partially hydrolyzed guar gum

SUMMARY:
The digestive process begins in the mouth and follows in the stomach and intestine. In the stomach the food is mixed with the gastric juices forming the chyme. To mix the food with the gastric juice as well as to provide gastric emptying (GE), the movements of the stomach are of great importance. Intestinal transit time is understood of the combination of GE, small intestine transit and colon transit time. The composition of the diet (lipid and protein content) exerts a direct influence on intestinal transit time due to the stimulation of hormone secretion, cholecystokinin and gastrin, respectively, which act to decrease GE velocity. In this context, it is also observed an important influence of dietary fibers on the speed of GE. Despite all knowledge about dietary fibers, information on such compounds still has many controversies. Due to the difficulty of finding compounds that fit into only one specific category (viscous, fermentable or prebiotic) there is difficulty in establishing a concept that best defines what are dietary fibers. The CODEX Alimentarius Commission in 2009 defined dietary fibers as carbohydrate polymers composed of ten or more monomer units of this macronutrient, which are not hydrolyzed by enzymes in the human intestine. Dietary fibers can be classified into insoluble and soluble according to the ability to bind to water molecules and form gels. Soluble fibers, especially those classified as prebiotic, in the intestine are fermented by bacteria giving rise to short chain fatty acids (SCFA). The SCFA stimulates the production and secretion of PYY and GLP-1 are associated with inhibition of gastric motility. Due to the importance of knowing the intestinal transit time, several methods have been developed, but scintigraphy is the gold standard technique for this analysis. Given the above and controversies present in the literature on the dietary fibers, there was a shortage of studies with the objective of evaluating the impact of different dietary fibers in intestinal transit time. This study shows relevant to help elucidate the behavior of different dietary fibers in intestinal transit time, offering data for correct and safe use of dietary fibers in various clinical situations. The hypothesis of this study is that the partially hydrolyzed guar gum delays the time of gastric emptying and intestinal transit, being this effect not observed for fructooligosaccharide

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers;
* Both sexes;
* Age Range:From 18 to 40 years old
* Volunteers who do not have gluten or egg restriction
* No history or diagnosis of gastrointestinal diseases;
* Had not undergone recent operations that compromised intestinal transit time and / or gastric emptying.

Exclusion Criteria:

* Volunteers who used prebiotic, probiotic and / or symbiotic volunteers at least 10 days prior to study day;
* Volunteers diagnosed with hypothyroidism and / or diabetes or who reported hypoglycemia and not tolerance to fasting;
* Women were asked about pregnancy, suspected pregnancy, use of contraceptive methods and menstrual cycle. If there was any possibility of pregnancy, based on these questions, the volunteer was excluded from the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-07-21 (Actual); Primary Completion 2019-04-13 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Gastric Emptying Time and intestinal transit time | After the 3rd day of the protocol
  The impact of the fibers under the gastric emptying and intestinal transit time is evaluated after the volunteer performs the ingestion of the 3 modules on different days.

SECONDARY OUTCOMES:
Intestinal Hormones Concentrations | Up to 3 weeks after protocol termination
  Dosage of serum concentrations
Compare gastric emptying and intestinal transit times between dietary fiber types | Up to 3 weeks after protocol termination
  To compare how the fibers influenced the time of gastric emptying and intestinal transit

CONTACTS AND LOCATIONS:
Overall Officials: Simone V Generoso, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Escola de Enfermagem - UFMG, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No